CLINICAL TRIAL: NCT05457647
Title: Assessment of Theranostic Guided Riboflavin/UV-A Corneal Cross-linking for Treatment of Keratoconus
Brief Title: Theranostic Guided Riboflavin/UV-A Corneal Cross-linking
Acronym: ARGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regensight (Industry)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RSKC001
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Keratoconus
Keywords: theranostics; riboflavin; UV-A light; corneal cross-linking
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Intervention Model Description: One study arm receiving riboflavin/UV-A corneal cross-linking with either standard, epi-off, or transepithelial, epi-on, treatment protocol. Only one eye of each participant is designated as the study eye. If both eyes of a study participant are eligible, the eye with worst CDVA is enrolled and treated.
Masking Description: Outcome assessor is masked. Statistician is masked. Participant receives stratification to either corneal cross-linking protocol after consent form signature.
  All participants wear contact lens after treatment until first postoperative eye examination at 1 week, when the corneal epithelium is completely healed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Riboflavin/UV-A corneal cross-linking monitored by theranostic software module (Experimental): One study arm receiving riboflavin/UV-A corneal cross-linking with either standard, epi-off, or transepithelial, epi-on, treatment protocol. Only one eye of each participant is designated as the study eye.
  Interventions: Device: Riboflavin/UV-A corneal cross-linking

INTERVENTIONS:
Device: Riboflavin/UV-A corneal cross-linking — Corneal cross-linking procedure is performed using the C4V CHROMO4VIS™ medical device equipped with theranostic software module in all participants. Participants will receive a single dose of the 0.22% riboflavin ophthalmic solution, RitSight™. Application of the riboflavin eye drop is done for 15 minutes for the epi-off CXL treatment and 20 minutes for the epi-on CXL treatment. Estimates of riboflavin concentration into the cornea are monitored by the C4V CHROMO4VIS™ system during the dosing phase of treatment. Once the pre-set dosing phase is completed, the C4V CHROMO4VIS™ system provides the Operator the access to the UV-A light irradiation of the cornea with 5.4 J/cm2 total energy dose (10 mW/cm2 for 9 min.) and 7.00 mm light beam diameter in all participants. Estimates of treatment efficacy by calculation of theranostic score are performed by the C4V CHROMO4VIS™ system during UV-A light irradiation.

SUMMARY:
This is a clinical study consisting of a study arm to validate accuracy and precision of the combined use of theranostic imaging biomarkers, riboflavin score and theranostic score, to assess and predict efficacy of corneal cross-linking in flattening the corneal topography Kmax value at 12-months postoperatively. The objective of the study is to assess the performance of the theranostic software module (Research Use Only) of a CE marked (CE1936) UV-A medical device, C4V CHROMO4VIS™, in order to validate its use for theranostic-guided corneal cross-linking treatment of keratoconus and corneal ectasia. The study hypothesis is that theranostic-guided riboflavin/UV-A corneal cross-linking with the C4V CHROMO4VIS™ system is safe and can estimate treatment efficacy during operation, regardless of treatment protocol, i.e., either with or without epithelial removal.

DETAILED DESCRIPTION:
Keratoconus is a naturally-occurring ocular condition characterized by progressive thinning and steepening of the central cornea, resulting in corneal optical irregularities with increasing myopia, irregular astigmatism, corneal opacity and consequential loss of visual acuity. Riboflavin/UV-A corneal cross-linking is a procedure used to biomechanically stabilize the weak cornea in keratoconus and to slow down or halt the clinical progression of this disease. Theranostics is an emerging therapeutic paradigm that enables monitoring of image-guided therapy through the use of a theranostic module that makes use of real-time non-invasive molecular imaging analysis of the tissue being treated to achieve optimal treatment outcomes in the management of disease on a personal basis.

The theranostic software module of the C4V CHROMO4VIS™ medical device is able to measure the concentration of riboflavin into the cornea during treatment (i.e., the riboflavin score) and to provide the surgeon with an objective assessment of treatment efficacy (i.e., the theranostic score).

The scope of this study is to validate the combined use of the theranostic imaging biomarkers in predicting the flattening of corneal topography Kmax value at 1-year postoperatively. The 1-year follow-up is long enough to provide scientific evidence of the safety and efficacy of the theranostic UV-A medical device in question. A pre-operative examination ensures that every interested and willing participant fulfils the inclusion criteria of this study. Masked post-operative examinations are carried out after 1 week, 1 month, 3 months, 6 months and 12 months.

This is a multi-center clinical trial. Eligible participants are stratified with allocation ratio 1:1 into either treatment protocol (epi-off CXL and epi-on CXL) using a computer-generated stratification plan with blocks. Two different blocks are created, which include eyes with Kmax steeper or flatter than 54.0 D to allocate patients with comparable baseline Kmax values in either treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

criteria for inclusion in the clinical trial are those currently referred to as the golden standard for the treatment of corneal cross-linking. The criterion to determine progression of keratoconus is based on providing at least one of the following evidences:

* at least two Placido disk corneal topography measurements showing at least +1.00 D steepening of the Kmax value in the last year or longer interval period.
* at least two manifest refraction measurements showing at least -0.50 D change in spherical equivalent refraction in the last year or longer interval period.
* at least two central corneal thickness (CCT) measurements showing at least -10 µm change in in the last year or longer interval period.

Exclusion Criteria:

* Anterior corneal curvature steeper than 63 D;
* Corneal thickness thinner than 400 µm;
* Corneal scarring;
* Descemetocele;
* History of herpetic keratitis;
* Concomitant eye diseases;
* Inflammatory eye diseases;
* Glaucoma;
* Cataract;
* Nistagmus;
* Pregnancy;
* Breast feeding.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Scorcia, MD, Principal Investigator — Azienda Ospedaliera Universitaria Mater Domini - Università Magna Graecia di Catanzaro; Marco Lombardo, MD, PhD, Study Director — Studio Italiano di Oftalmologia
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Universitaria Mater Domini - Università Magna Graecia di Catanzaro, Catanzaro
  - Azienda Ospedaliera Universitaria Careggi, Università di Firenze, Florence
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Università di Messina, Messina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lombardo G, Villari V, Micali NL, Leone N, Labate C, De Santo MP, Lombardo M. Non-invasive optical method for real-time assessment of intracorneal riboflavin concentration and efficacy of corneal cross-linking. J Biophotonics. 2018 Jul;11(7):e201800028. doi: 10.1002/jbio.201800028. Epub 2018 Apr 10. PMID 29451741
- [Background] Lombardo M, Lombardo G. Noninvasive real-time assessment of riboflavin consumption in standard and accelerated corneal crosslinking. J Cataract Refract Surg. 2019 Jan;45(1):80-86. doi: 10.1016/j.jcrs.2018.07.062. Epub 2018 Oct 22. PMID 30360937
- [Background] Lombardo G, Serrao S, Lombardo M. Comparison between standard and transepithelial corneal crosslinking using a theranostic UV-A device. Graefes Arch Clin Exp Ophthalmol. 2020 Apr;258(4):829-834. doi: 10.1007/s00417-019-04595-6. Epub 2020 Jan 3. PMID 31900647
- [Background] Lombardo G, Micali NL, Villari V, Serrao S, Lombardo M. All-Optical Method to Assess Stromal Concentration of Riboflavin in Conventional and Accelerated UV-A Irradiation of the Human Cornea. Invest Ophthalmol Vis Sci. 2016 Feb;57(2):476-83. doi: 10.1167/iovs.15-18651. PMID 26868750
- [Background] Lombardo M, Pucci G, Barberi R, Lombardo G. Interaction of ultraviolet light with the cornea: clinical implications for corneal crosslinking. J Cataract Refract Surg. 2015 Feb;41(2):446-59. doi: 10.1016/j.jcrs.2014.12.013. Epub 2014 Dec 23. PMID 25542349
- [Background] Lombardo G, Bernava GM, Serrao S, Lombardo M. Theranostic-guided corneal cross-linking: Preclinical evidence on a new treatment paradigm for keratoconus. J Biophotonics. 2022 Dec;15(12):e202200218. doi: 10.1002/jbio.202200218. Epub 2022 Sep 16. PMID 36059083
- [Background] Roszkowska AM, Lombardo G, Mencucci R, Scorcia V, Giannaccare G, Vestri A, Alunni Fegatelli D, Bernava GM, Serrao S, Lombardo M. A randomized clinical trial assessing theranostic-guided corneal cross-linking for treating keratoconus: the ARGO protocol. Int Ophthalmol. 2023 Jul;43(7):2315-2328. doi: 10.1007/s10792-022-02628-4. Epub 2022 Dec 31. PMID 36587174
- [Result] Roszkowska AM, Scorcia V, Mencucci R, Giannaccare G, Lombardo G, Alunni Fegatelli D, Vestri A, Bifezzi L, Bernava GM, Serrao S, Lombardo M. Assessment of the Predictive Ability of Theranostics for Corneal Cross-linking in Treating Keratoconus: A Randomized Clinical Trial. Ophthalmology. 2024 Dec;131(12):1403-1415. doi: 10.1016/j.ophtha.2024.06.012. Epub 2024 Jun 20. PMID 38908553
- See also: Updates on clinical trial RSKC001 — https://regensight.com/en/science-technology/

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module: One study arm receiving riboflavin/UV-A corneal cross-linking with either standard, Epi-OFF, or transepithelial, Epi-ON, treatment protocol. Only one eye of each participant is designated as the study eye.
  Riboflavin/UV-A corneal cross-linking: Corneal cross-linking procedure is performed using the C4V CHROMO4VIS™ system equipped with theranostic software module in all participants. Participants will receive a single dose of the 0.22% riboflavin ophthalmic solution, RitSight™. Application of the riboflavin eye drop is done for 15 minutes for the EpiOFF CXL treatment and 20 minutes for the EpiON CXL treatment. Estimates of riboflavin concentration into the cornea are monitored by the C4V CHROMO4VIS™ system during the dosing phase of treatment. Once the pre-set dosing phase is completed, the C4V CHROMO4VIS™ system provides the Operator the access to the UV-A irradiation of the cornea with 5.4 J/cm2 total energy dose (10 mW/cm2 for 9 min.) and 7.00 mm light beam diameter in all participants. Estimates of treatment efficacy by calculation of theranostic score are performed by the C4V CHROMO4VIS™ system during UV-A irradiation.
Period: Overall Study
Arm/Group | Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module
Started | 50; 50 eyes
Completed | 47; 47 eyes
Not Completed | 3; 3 eyes
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Participants had confirmed diagnosis of progressive keratoconus using Placido disc corneal topography
Arm/Group | Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 50
Medical history [Number; unit: participants]
  Positive family history of keratoconus | 12
  History of allergy/dermatitis | 4
  History of hypothyroidism | 3
  History of diabetes mellitus | 1
  History of systemic lupus erythematosus and ulcerative colitis | 1

OUTCOME MEASURES:

1. Primary Outcome: Validation of the Theranostic Scores
Description: The aim of this study is to validate the combined use of theranostic imaging biomarkers in predicting the propsensity of corneal corneal cross-linking (CXL) in flattening the Kmax at 1-year.
  The accuracy and precision (95% CI) of the combined use of the theranostic imaging biomarkers to predict CXL treatment outcome are determined by calculating the percentage of correctly classified eyes and the positive predictive value (PPV) respectively.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Percentage
Units Other Than Participants: Eyes
Arm/Group | Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module
Number analyzed (Participants) | 47
Number analyzed (Eyes) | 47
Percentage
  Accuracy | 91 [79 to 98]
  Precision | 95 [89 to 99]
Statistical Analysis 1: Comparison: Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module; Accuracy and precision of the combined use of theranostic imaging biomarkers generated by the UV-A device to predict the propensity of CXL in flattening the Kmax value at 12-months; Test type: Other — The accuracy and precision of the theranostic imaging biomarkers, including both the riboflavin score and theranostic score, to predict CXL treatment outcome were determined by calculating the proportion of correctly classified eyes and the positive predictive value respectively; Proportion = 91 — The study set a minimum threshold of 85 for the the combined use of the theranostic imaging biomarkers' accuracy and precision in predicting the propensity of CXL to halt disease progression at 1 year in the study population

2. Secondary Outcome: Corneal Topography
Description: Change of Maximum Keratometry value of Placido disc corneal topography. The secondary outcome measure of efficacy was assessed by measuring changes of Kmax value (D) from baseline to 12 months postoperatively.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: Eyes
Groups:
- Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module: One study arm receiving riboflavin/UV-A corneal cross-linking with either standard, epi-off, or transepithelial, epi-on, treatment protocol. Only one eye of each participant is designated as the study eye.
  Riboflavin/UV-A corneal cross-linking: corneal cross-linking procedure is performed using the C4V CHROMO4VIS™ system equipped with theranostic software module in all participants. Participants will receive a single dose of the 0.22% riboflavin ophthalmic solution, RitSight™. Application of the riboflavin eye drop is done for 15 minutes for the epi-off CXL treatment and 20 minutes for the epi-on CXL treatment. Estimates of riboflavin concentration into the cornea are monitored by the C4V CHROMO4VIS™ system during the dosing phase of treatment. Once the pre-set dosing phase is completed, the C4V CHROMO4VIS™ system provides the Operator the access to the UV-A irradiation of the cornea with 5.4 J/cm2 total energy dose (10 mW/cm2 for 9 min.) and 7.00 mm light beam diameter in all participants. Estimates of treatment efficacy by calculation of theranostic score are performed by the C4V CHROMO4VIS™ system during UV-A irradiation.
Arm/Group | Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module
Number analyzed (Participants) | 47
Number analyzed (Eyes) | 47
diopters | -1.5 (1.6)
Statistical Analysis 1: Comparison: Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module; Assessment of change of Kmax value at 12-months follow-up visit; Test type: Other — Paired Wilcoxon signed-rank test was used to compare the distributions preoperatively and 12-months postoperatively; p < 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Endothelial Cell Density
Description: Change of Endothelial Cell Density (ECD) of the cornea. The secondary outcome measure of safety was assessed by measuring change of ECD (cell/mm^2) from baseline to 12 months postoperatively.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cells/mm^2
Units Other Than Participants: Eyes
Arm/Group | Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module
Number analyzed (Participants) | 47
Number analyzed (Eyes) | 47
cells/mm^2 | -63 (336)
Statistical Analysis 1: Comparison: Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module; Assessment of change of ECD value at 12-months follow-up visit; Test type: Other — Paired Wilcoxon signed-rank test was used to compare the distributions preoperatively and 12-months postoperatively; p < 0.05, Wilcoxon (Mann-Whitney)

4. Other Pre Specified Outcome: Manifest Refraction
Description: Change of Manifest Spherical Equivalent Refraction (MSER). This outcome was assessed by measuring change of MSER (D) from baseline to 12 months postoperatively.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module
Number analyzed (Participants) | 47
diopters | 0.2 (1.2)
Statistical Analysis 1: Comparison: Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module; Assessment of change of MSER value at 12-months follow-up visit; Test type: Other — Paired Wilcoxon signed-rank test was used to compare the distributions preoperatively and 12-months postoperatively; p < 0.05, Wilcoxon (Mann-Whitney)

5. Other Pre Specified Outcome: Corrected Distance Visual Acuity
Description: Change of Corrected Distance Visual Acuity (CDVA) measured with ETDRS chart and expressed in LogMAR.
  This outcome was assessed by measuring changes of CDVA from baseline to 12 months postoperatively.
  A negative change means improvement in CDVA after treatment.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module
Number analyzed (Participants) | 47
Number analyzed (Eyes) | 47
LogMAR | -0.1 (0.1)
Statistical Analysis 1: Comparison: Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module; Assessment of change of CDVA value at 12-months follow-up visit; Test type: Other — Paired Wilcoxon signed-rank test was used to compare the distributions preoperatively and 12-months postoperatively; p < 0.05, Wilcoxon (Mann-Whitney)

6. Other Pre Specified Outcome: Uncorrected Distance Visual Acuity
Description: Change of Uncorrected Distance Visual Acuity (UDVA) measured with ETDRS chart and expressed in LogMAR.
  This outcome was assessed by measuring changes of UDVA from baseline to 12 months postoperatively.
  A negative change means improvement in UDVA after treatment.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module
Number analyzed (Participants) | 47
Number analyzed (Eyes) | 47
LogMAR | -0.1 (0.1)
Statistical Analysis 1: Comparison: Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module; Assessment of change of UDVA value at 12-months follow-up visit; Test type: Other — Paired Wilcoxon signed-rank test was used to compare the distributions preoperatively and 12-months postoperatively; p < 0.05, Wilcoxon (Mann-Whitney)

7. Other Pre Specified Outcome: Central Corneal Thickness
Description: Change of Central Corneal Thickness (CCT). This outcome was assessed by measuring changes of CCT from baseline to 12 months postoperatively.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: micrometers
Units Other Than Participants: Eyes
Arm/Group | Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module
Number analyzed (Participants) | 47
Number analyzed (Eyes) | 47
micrometers | -5 (18)
Statistical Analysis 1: Comparison: Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module; Assessment of change of CCT value at 12-months follow-up visit; Test type: Other — Paired Wilcoxon signed-rank test was used to compare the distributions preoperatively and 12-months postoperatively; p < 0.05, Wilcoxon (Mann-Whitney)

8. Other Pre Specified Outcome: Stratification Groups
Description: Change of primary and secondary outcome measures in either stratification group (epi-off CXL protocol and epi-on CXL protocol).
  These exploratory outcome measures included the following assessment: assessmentg of changes of Kmax value (D) at 12-months postoperatively in either stratification group.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: diopters
Units Other Than Participants: Eyes
Groups:
- Epi-off Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module: Stratification arm receiving riboflavin/UV-A corneal cross-linking with epi-off treatment protocol. Only one eye of each participant is designated as the study eye.
  Participants receive a single dose of the 0.22% riboflavin ophthalmic solution, RitSight™. Application of the riboflavin eye drop is done for 15 minutes for the epi-off CXL treatment. Estimates of riboflavin concentration into the cornea are monitored by the C4V CHROMO4VIS™ system during the dosing phase of treatment. Once the pre-set dosing phase is completed, the C4V CHROMO4VIS™ system provides the Operator the access to the UV-A irradiation of the cornea with 5.4 J/cm2 total energy dose (10 mW/cm2 for 9 min.) and 7.00 mm light beam diameter in all participants. Estimates of treatment efficacy by calculation of theranostic score are performed by the C4V CHROMO4VIS™ system during UV-A irradiation.
- Epi-on Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module: Stratification arm receiving riboflavin/UV-A corneal cross-linking with epi-on treatment protocol. Only one eye of each participant is designated as the study eye.
  Participants receive a single dose of the 0.22% riboflavin ophthalmic solution, RitSight™. Application of the riboflavin eye drop is done for 20 minutes for the epi-on CXL treatment. Estimates of riboflavin concentration into the cornea are monitored by the C4V CHROMO4VIS™ system during the dosing phase of treatment. Once the pre-set dosing phase is completed, the C4V CHROMO4VIS™ system provides the Operator the access to the UV-A irradiation of the cornea with 5.4 J/cm2 total energy dose (10 mW/cm2 for 9 min.) and 7.00 mm light beam diameter in all participants. Estimates of treatment efficacy by calculation of theranostic score are performed by the C4V CHROMO4VIS™ system during UV-A irradiation.
Arm/Group | Epi-off Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module | Epi-on Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module
Number analyzed (Participants) | 24 | 23
Number analyzed (Eyes) | 24 | 23
diopters | -1.9 (2.0) | -1.1 (1.0)
Statistical Analysis 1: Comparison: Epi-off Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module vs Epi-on Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module; Test type: Other — Paired Wilcoxon signed-rank test was used to compare the distributions preoperatively and 12-months postoperatively. Bonferroni correction was applied to analysis of exploratory outcome measures of stratification groups; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1-week, 1-month, 3-months, 6-months and 12-months,.
Description: Corneal haze was the only adverse events recorded.
Arm/Group | Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 6/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Riboflavin/UV-A Corneal Cross-linking Monitored by Theranostic Software Module (N=50)
Corneal Haze (Eye disorders) | 6 — Frequency of corneal haze was maximum at 1 month

LIMITATIONS AND CAVEATS:
This study assessed CXL efficacy by measuring the change of the Kmax index, which was aligned with commonly used approaches in the field.

The list of adverse events may not be fully comprehensive as the first postoperative visit was scheduled at 7 days after treatment, excluding immediate postoperative events, such as eye pain, stromal oedema, corneal striae and conjunctival hyperaemia, from the assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT05457647/Prot_SAP_000.pdf